CLINICAL TRIAL: NCT04937647
Title: Collection of Endoscopic Images and Videos for Validation of Artificial Intelligence Algorithms for Computer Aided Detection and Characterisation of Early Gastrointestinal Neoplasia
Brief Title: Evaluation of Neoplasia With Artificial Intelligence in Gastrointestinal Endoscopy
Acronym: NEW-AGE
Status: Recruiting | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2020/58
Record Dates: First submitted 2021-06-09; First posted 2021-06-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Neoplasms
Keywords: gastrointestinal neoplasia; artificial intelligence
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Videotape Recording

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: collection of endoscopic images and videos — collection of endoscopic images and videos

SUMMARY:
This study aims to validate and evaluate AI algorithms for detection and characterization of early GI neoplasia.

DETAILED DESCRIPTION:
This is an investigator initiated; multi-centre study and will be conducted in two phases. Validation & Optimization phase, where routinely collected and anonymized endoscopic images and videos from the departmental teaching and training library will be used to validate, and if needed fine-tune and improve, the accuracy of an AI algorithm. Testing phase, where the evaluation of AI algorithms performance will be conducted on a prospective basis. The ground truth (standard) will be expert assessment and histological diagnosis.

This study has no direct impact on patient's clinical care, and collection of all endoscopic data will take place during standard endoscopy procedures done for purely clinical indications. No additional procedures, biopsies or interventions will be performed as a part of this study.

ELIGIBILITY:
Inclusion Criteria:

-The participant must meet ALL of the following criteria to be considered eligible for the study:

* Male or Female, aged 18 years or above.
* Requiring gastroscopy and/or colonoscopy to investigate gastrointestinal symptoms, or as part of screening or ongoing surveillance of GI neoplasia.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria

The participant may not enter the study if ANY of the following apply:

* Patients with endoscopically active severe oesophagitis
* Poor bowel preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In phase (1), all previously collected, anonymized and stored endoscopic images and videos of early GI neoplasia in the departmental endoscopy teaching and training library. In phase (2), all eligible patients coming for upper and/or lower GI endoscopy for clinical reasons in participating centres will be approached for enrolment into this study.
Sampling Method: Probability Sample
Enrollment: 1650 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
neoplasia detection rate | during the procedure, up to 24 weeks, at 1 year, through study completion
  neoplasia detection rate of the AI algorithms in different locations of the GI tract.

SECONDARY OUTCOMES:
Accuracy of AI diagnosis | during the procedure, up to 24 weeks, at 1 year, through study completion
  Accuracy of real time optical diagnosis (characterization) of GI neoplasia by the AI algorithm.
Endoscopist neoplasia detection rate | during the procedure, up to 24 weeks, at 1 year, through study completion
  Detection rate of endoscopists at various levels of experience

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Bhandari, Prof, Principal Investigator — Portsmouth Hospitals University NHS Trust
Locations (1):
- Portsmouth Hospitals NHS University Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No